CLINICAL TRIAL: NCT01129440
Title: Glass Ionomer Sealant and Fluoride Varnish Randomized Clinical Trial
Brief Title: Glass Ionomer Sealant and Fluoride Varnish Study to Prevent Early Childhood Caries
Acronym: GIFVT
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: National Institute of Dental and Craniofacial Research (NIDCR) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: NIDCR 09-014-E; U54DE019285 (NIH)
Record Dates: First submitted 2010-05-21; First posted 2010-05-24 (Estimated); Results first posted 2020-02-19 (Actual); Last update posted 2020-03-04 (Actual); Status verified 2020-02

CONDITIONS: Dental Caries
Keywords: Children; Fluoride varnish; Glass ionomer sealant; Prevention
MeSH Terms: conditions — Dental Caries

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Fluoride Varnish (Active Comparator): Topical fluoride varnish (FV) applications every 6 months
  Interventions: Device: Fluoride Varnish
- FV + Glass Ionomer Sealants (Experimental): Topical fluoride varnish (FV) applications every 6 months, and fluoride-releasing glass ionomer sealants (GIS) placed on primary molars at baseline and annually, as needed
  Interventions: Device: Fluoride Varnish; Device: Glass Ionomer Sealant

INTERVENTIONS:
Device: Fluoride Varnish — Topical application of 0.25mL of fluoride varnish on each dental arch (upper and lower) at baseline and every 6 months.
  Other Names: 3M ESPE CavityShield® single-dose fluoride varnish units
Device: Glass Ionomer Sealant — Fluoroaluminosilicate glass powder and polyacrylic acid liquid are mixed together in a capsule to form the glass ionomer sealant material.
  After toothbrushing and conditioning dental surfaces with 20% polyacrylic acid for 10 seconds, pink-colored fluoride releasing glass ionomer dispensed from a capsule is applied to the occlusal (biting) surface of the molar.
  Other Names: GC Fuji TRIAGE CAPSULE and its conditioner
  Arms: FV + Glass Ionomer Sealants

SUMMARY:
The goal of this project is to conduct a community-based randomized clinical trial to compare the caries prevention efficacy of fluoride varnish applied every six months vs. fluoride varnish applied every six months and fluoride releasing glass ionomer sealants applied annually to the eligible occlusal surfaces of primary molars in 3-6-year-old children.

DETAILED DESCRIPTION:
Community-based, stratified (by location) randomized clinical trial (RCT) to determine the relative efficacy of topically applied fluoride varnish (FV) applications alone vs FV with fluoride-releasing glass ionomer (GI) sealants on occlusal surfaces of primary molars in reducing the caries incidence and increment in 3-6 year old children. A parallel groups design RCT stratified by study site (one dental and one non-dental location) will be conducted among 596 initially 2.5- to 3-year-old children. Those eligible will be randomized to one of 2 groups (FV or GIS+FV) and followed for 36 months. The RCT will take place at two sites serving primarily underserved, minority and low-income populations in Southern California: 1) the dental facility of the San Ysidro Health Center (SYHC) located near the U.S.-Mexican Border serves mainly Latino immigrants, and 2) the Comprehensive Health Center - Ocean View (CHC-OV), in a non-dental setting in close proximity to its dental clinic, which serves Latinos and African Americans. Both sites are part of a consortium of community clinics (SYHC Inc) and are located 15 miles apart from each other.

Annual study dental examinations will be performed by trained, calibrated, study dentists to determine caries (precavitated and cavitated) incidence and increment. Children identified as needing dental care will be referred for appropriate treatment.

ELIGIBILITY:
Inclusion Criteria:

* Family resides in the South Bay or Central San Diego area
* Parent/Guardian can consent in English or Spanish
* Child has 1-8 caries-free primary molars (with no occlusal pre-cavitation and no restoration)
* Child is cooperative and behaviorally suited for the clinical trial interventions
* Child is a registered patient at San Ysidro Health Center Inc.

Exclusion Criteria:

* Any siblings of participants
* Child with cavitated lesions
* Child with a health condition, special need, or with a complicated factor that will prevent from completing the required number of visits during a 36-month follow-up period
* Anything, that in the opinion of the investigator, would preclude the child from complying with the protocol or jeopardize the safety of the child while on the protocol

Ages: 2 Years to 3 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 597 (Actual)
Dates: Start 2011-06; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Francisco Ramos-Gomez, DDS, MS, MPH, Principal Investigator — University of California, Los Angeles; Stuart Gansky, DrPH, Principal Investigator — University of California, San Francisco
Locations (1):
- San Ysidro Health Center, San Ysidro, California, United States

IPD SHARING:
Plan to Share IPD: Yes
UCSF DataShare (http://datashare.ucsf.edu) is no longer functional. The Data Dryad repository (https://datadryad.org) will be utilized instead.

REFERENCES:
- [Result] Garcia RI, Gregorich SE, Ramos-Gomez F, Braun PA, Wilson A, Albino J, Tiwari T, Harper M, Batliner TS, Rasmussen M, Cheng NF, Santo W, Geltman PL, Henshaw M, Gansky SA. Absence of Fluoride Varnish-Related Adverse Events in Caries Prevention Trials in Young Children, United States. Prev Chronic Dis. 2017 Feb 16;14:E17. doi: 10.5888/pcd14.160372. PMID 28207379
- [Result] Tiwari T, Casciello A, Gansky SA, Henshaw M, Ramos-Gomez F, Rasmussen M, Garcia RI, Albino J, Batliner TS; Early Childhood Caries Collaborating Centers. Recruitment for health disparities preventive intervention trials: the early childhood caries collaborating centers. Prev Chronic Dis. 2014 Aug 7;11:E133. doi: 10.5888/pcd11.140140. PMID 25101490
- [Result] Garcia RI, Tiwari T, Ramos-Gomez F, Heaton B, Orozco M, Rasmussen M, Braun P, Henshaw M, Borrelli B, Albino J, Diamond C, Gebel C, Batliner TS, Barker JC, Gregorich S, Gansky SA. Retention strategies for health disparities preventive trials: findings from the Early Childhood Caries Collaborating Centers. J Public Health Dent. 2017 Dec;77(1):63-77. doi: 10.1111/jphd.12182. Epub 2016 Oct 19. PMID 27759164
- [Derived] Albino J, Tiwari T, Gansky SA, Henshaw MM, Barker JC, Brega AG, Gregorich SE, Heaton B, Batliner TS, Borrelli B, Geltman P, Kressin NR, Weintraub JA, Finlayson TL, Garcia RI; Early Childhood Caries Collaborating Centers. The basic research factors questionnaire for studying early childhood caries. BMC Oral Health. 2017 May 19;17(1):83. doi: 10.1186/s12903-017-0374-5. PMID 28526003

RESULTS

PARTICIPANT FLOW:
Groups:
- FV + Glass Ionomer Sealants: Topical fluoride varnish (FV) applications every 6 months, and fluoride-releasing glass ionomer sealants (GIS) placed on primary molars at baseline and annually, as needed
  Fluoride Varnish: Topical application of 0.25mL of fluoride varnish on each dental arch (upper and lower) at baseline and every 6 months.
  Glass Ionomer Sealant: Fluoroaluminosilicate glass powder and polyacrylic acid liquid are mixed together in a capsule to form the glass ionomer sealant material.
  After toothbrushing and conditioning dental surfaces with 20% polyacrylic acid for 10 seconds, pink-colored fluoride releasing glass ionomer dispensed from a capsule is applied to the occlusal (biting) surface of the molar.
Period: Overall Study
Arm/Group | Fluoride Varnish | FV + Glass Ionomer Sealants
Started | 297 | 300
12 Month Follow-up | 249 | 256
24 Month Follow-up | 239 | 258
Completed | 246 | 258
Not Completed | 51 | 42

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Fluoride Varnish | FV + Glass Ionomer Sealants | Total
Number analyzed (Participants) | 297 | 300 | 597
Age, Continuous [Mean (Standard Deviation); unit: years] | 3.4 (0.43) | 3.4 (0.48) | 3.4 (0.46)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 166 | 154 | 320
  Male | 131 | 146 | 277
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 288 | 284 | 572
  Not Hispanic or Latino | 9 | 13 | 22
  Unknown or Not Reported | 0 | 3 | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 6 | 8 | 14
  White | 289 | 285 | 574
  More than one race | 0 | 3 | 3
  Unknown or Not Reported | 1 | 4 | 5
Center [Count of Participants; unit: Participants]
  Center 1 | 148 | 151 | 299
  Center 2 | 149 | 149 | 298

OUTCOME MEASURES:

1. Primary Outcome: Caries Incidence
Description: Caries incidence by 36 months measured by whether the change in the number of decayed, missing, or filled primary tooth surfaces (dmfs) index increased from baseline (ie. change in dmfs >0)
Time Frame: Assessed every 12 months (plus or minus 1 month); Month 36 reported
Measure: Count of Participants; unit: Participants
Arm/Group | Fluoride Varnish | FV + Glass Ionomer Sealants
Number analyzed (Participants) | 246 | 258
Participants | 137 | 123

2. Primary Outcome: Caries Increment
Description: Caries increment by 36 months measured by the amount of change in dmfs index from baseline
Time Frame: Assessed every 12 months (plus or minus 1 month); Month 36 reported
Measure: Mean (95% Confidence Interval); unit: tooth surfaces
Arm/Group | Fluoride Varnish | FV + Glass Ionomer Sealants
Number analyzed (Participants) | 246 | 258
tooth surfaces | 4.9 [4.0 to 5.9] | 4.1 [3.3 to 5.0]

3. Secondary Outcome: Caries Patterns
Description: Determine and compare caries patterns (maxillary incisor smooth surfaces, posterior occlusal surfaces) across study arms over time.
  Occlusal surface dmfs>0 in baseline eligible molar teeth.
Time Frame: Assessed every 12 months (plus or minus 1 month); Month 36 reported
Measure: Count of Participants; unit: Participants
Arm/Group | Fluoride Varnish | FV + Glass Ionomer Sealants
Number analyzed (Participants) | 246 | 258
Participants | 117 | 106

4. Secondary Outcome: Salivary Fluoride Level
Description: Relative changes in salivary fluoride levels pre- and post-treatment will be measured from a subsample of participating children
Time Frame: Every 6 months (plus minus 1 month); Month 30 reported
Population: Randomly selected subset with salivary fluoride measured
Measure: Mean (Standard Deviation); unit: ppm
Arm/Group | Fluoride Varnish | FV + Glass Ionomer Sealants
Number analyzed (Participants) | 35 | 34
ppm | 0.072 (0.108) | 0.128 (0.494)

5. Secondary Outcome: Retention of Glass Ionomer Sealants
Description: Retention and maintenance of fluoride-releasing glass ionomer sealants will be recorded from a subset of children using an intraoral digital camera
Time Frame: Assessed every at 12 months and 24 months (plus minus 1 month); Month 24 reported
Measure: Count of Participants; unit: Participants
Arm/Group | FV + Glass Ionomer Sealants
Number analyzed (Participants) | 265
Participants | 249

6. Secondary Outcome: Adverse Event
Description: Clinician mediated adverse event up to 7 days after fluoride varnish application, ascertained through follow-up telephone call 5-14 days after application.
Time Frame: every 6 months; up to 7 days after application
Measure: Count of Participants; unit: Participants
Arm/Group | Fluoride Varnish | FV + Glass Ionomer Sealants
Number analyzed (Participants) | 297 | 300
Participants | 0 | 1

7. Other Pre Specified Outcome: Effect Modification of Caries Incidence and Increment by Location
Description: Caries increment measured by the amount of change in dmfs index from baseline separately by location and caries incidence measured by whether the change in dmfs index increased (ie. change in dmfs >0) separately by location.
  Subgroup analyses will be performed with statistical models which have the location, the intervention group, and their interaction to assess possible effect modification (i.e. moderation).
Time Frame: Assessed every 12 months (plus minus 1 month)
Reporting Status: Not Posted

8. Other Pre Specified Outcome: Effect Modification of Caries Incidence and Increment by Baseline Frankl Child Behavior Score
Description: Caries increment measured by the amount of change in dmfs index from baseline separately by baseline Frankl child behavior score and caries incidence measured by whether the change in dmfs index increased (ie. change in dmfs >0) separately by Frankl score.
  Subgroup analyses will be performed with statistical models which have the baseline Frankl score, the intervention group, and their interaction to assess possible effect modification (i.e. moderation).
Time Frame: Assessed every 12 months (plus minus 1 month)
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 36 months
Arm/Group | Fluoride Varnish | FV + Glass Ionomer Sealants
All-Cause Mortality (participants affected / at risk) | 0/297 | 0/300
Serious Adverse Events (participants affected / at risk) | 0/297 | 0/300
Other Adverse Events (participants affected / at risk) | 0/297 | 1/300
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Fluoride Varnish (N=297) | FV + Glass Ionomer Sealants (N=300)
Viral infection (Infections and infestations) | 0 | 1 — Fever that a physician diagnosed as a viral infection. Study team judged AE as unrelated to study intervention and DSMB concurred. Garcia et al. 2017, PMC5313125.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No